CLINICAL TRIAL: NCT01461109
Title: Evaluation of [18F] CFPyPB PET as a Marker of Glycine Transporter-1 (GlyT1) Receptor in Subjects With Parkinson Disease, Alzheimer Disease and Healthy Subjects
Brief Title: Research Involving Subjects With Parkinson's Disease, Alzheimer Disease and Healthy Controls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Principal Investigator, David Russell, MD, PhD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GlyT1-01
Record Dates: First submitted 2011-09-27; First posted 2011-10-27 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Parkinson Disease; Alzheimer Disease
Keywords: Parkinson Disease; Alzheimer Disease; [18F] CFPyPB; GlyT1
MeSH Terms: conditions — Parkinson Disease; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assess [18F] CFPyPB and PET imaging (Experimental): To assess [18F]CFPyPB and PET imaging
  Interventions: Drug: [18F] CFPyPB

INTERVENTIONS:
Drug: [18F] CFPyPB — Each subject will receive a bolus injection targeted to be 5 mCi and not to exceed 5.5 mCi (not >10% of 5 mCi limit) of [18F]CFPyPB or 5 μg of CFPyPB (whichever is greatest).

SUMMARY:
The underlying goal of this study is to assess [18F] CFPyPB PET imaging as a tool to evaluate the activity of the GlyT1 receptors in the brain of Parkinson's Disease (PD) and Alzheimer Disease (AD) research participants.

DETAILED DESCRIPTION:
Approximately 6 subjects with Parkinson disease, 6 subjects with Alzheimer disease and 20 healthy control subjects will be recruited to participate in this study. All subjects will undergo written informed consent and a screening evaluation including baseline clinical laboratory testing, a baseline physical and neurological evaluation and baseline cognitive evaluations. Subjects will be asked to undergo a bolus injection of [18F] CFPyPB followed by serial PET imaging scans and plasma sampling for measurement of [18F] CFPyPB in plasma (both protein bound and free) over a period of up to 4 hours. The imaging analyses will be performed by an image-processing specialist who will remain masked to the procedures employed with each imaging acquisition. The primary imaging outcome measure will be the brain regional distribution volumes expressed as a brain tissue to plasma ratio of the radioligand, [18F] CFPyPB. Time to the peak uptake and amplitude of the peak uptake will be evaluated for all brain regions and the results for the PD and AD subjects will be compared with the HC subjects.

At least 2 weeks following the initial imaging visit subjects (up to 2 PD subjects, up to 2 AD subjects and up to 5 HC subjects) may be asked to return for a second injection and scanning procedure to evaluate the reproducibility of the imaging measure using this procedure. Subjects may decline participation in the second scan. Subjects will be requested to return for this second scan until enough second scan data is collected to evaluate the imaging outcome measure for reproducibility.

ELIGIBILITY:
PD subject inclusion criteria:

* The participant is 30 years or older.
* Written informed consent is obtained.
* Participants have a diagnosis of PD (based on UK Brain Bank Criteria).
* Modified Hoehn and Yahr stage of 1 - 4.
* For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F] CFPyPB injection.

PD subject exclusion criteria:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion.
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* The subject has any contraindication to MRI examination, e.g. metal implants or phobia as determined by the onsite radiologist performing the scan.
* The subject is a pregnant or nursing mother

AD subject inclusion criteria:

* The participant is 50 years or older.
* Written informed consent is obtained.
* Participants have a clinical diagnosis of probable Alzheimer disease in accordance with the DSM-IV-TR and according to (NINCDS/ADRDA) criteria.
* Participants do not fulfill the ICC criteria for probable DLB, the NINDS-AIREN for probable vascular dementia, or the Neary [Neary, et al. 1998] criteria for FTD.
* Clinical Dementia Rating Scale score 0.5, 1 or 2.
* Modified Hachinski Ischemia Scale score of ≤ 4.
* Geriatric Depression Scale (GDS) ≤ 10.
* For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F] CFPyPB injection.

AD subject exclusion criteria:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion.
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* The subject has any contraindication to MRI examination, e.g. metal implants or phobia as determined by the onsite radiologist performing the scan.
* The subject is a pregnant or nursing mother.

Healthy volunteer inclusion criteria:

* The participant is 18 years or older.
* Written informed consent is obtained.
* Negative history of neurological or psychiatric illness based on evaluation by a research physician.
* For females, non-child bearing potential a negative urine or blood pregnancy test on day of [18F] CFPyPB injection.

Healthy volunteer exclusion criteria:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion.
* The subject has any contraindication to MRI examination, e.g. metal implants or phobia as determined by the onsite radiologist performing the scan.
* The subject is a pregnant or nursing mother.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To assess the dynamic uptake and washout of [18F] CFPyPB | Approximately 2 years
  To assess the dynamic uptake and washout of [18F] CFPyPB, an imaging tracer targeting the glycine transporter-1 (GlyT1) receptor in brain, using positron emission tomography (PET) in subjects with Parkinson disease (PD) Alzheimer disease (AD) and healthy controls (HC).

SECONDARY OUTCOMES:
Perform blood metabolite characterization of [18F] CFPyPB | Approximately 2 years
  To perform blood metabolite characterization of [18F] CFPyPB in subjects with PD, AD and HC to determine the nature of metabolites in assessment of [18F] CFPyPB as a single positron computed tomography (PET) brain imaging agent.
To obtain safety data | Approximately 2 years
  To acquire safety data following injection of [18F] CFPyPB
Obtain test/retest reproductibility | Approximately 2 years
  To obtain test/retest reproducibility of quantitative PET outcome measures with [18F] CFPyPB

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, MD, PhD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute_Neurodegenerative_Disorders, New Haven, Connecticut, United States

REFERENCES:
- See also: Institute for Neurodegenerative Disorders — http://www.indd.org